CLINICAL TRIAL: NCT01231633
Title: Comparative Study of Initial Ozurdex (Dexamethasone Implant) Versus Avastin (Bevacizumab) in the Treatment of Macular Edema Following Central Retinal Vein Occlusion (CRVO)
Brief Title: Comparison of Initial Ozurdex (Dexamethasone Implant) to Avastin (Bevacizumab) for Treatment of Macular Edema Caused by Central Retinal Vein Occlusion (CRVO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Long Island Vitreoretinal Consultants (Other)
Responsible Party: Principal Investigator, Vincent. A. Deramo, M.D., Prinicipal Investigator, Long Island Vitreoretinal Consultants
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IST CRVO 1118147
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Macular Edema; Central Retinal Vein Occlusion
Keywords: Macular Edema; Central Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Calcium Dobesilate; Dexamethasone; Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Subjects randomized to this arm will receive one initial treatment with Ozurdex then treated with Avastin if needed.
  Interventions: Drug: Ozurdex; Drug: Avastin
- Group 2 (Active Comparator): Subjects randomized to this arm will receive one initial treatment with Avastin then treated with Avastin if needed.
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: Ozurdex — Ozurdex, 0.7mg dexamethasone
  Other Names: Dexamethasone implant
  Arms: Group 1
Drug: Avastin — Formulated as a 1.25mg/0.05ml sterile solution given by intravitreal injection monthly as needed.
  Other Names: Avastin, bevacizumab

SUMMARY:
The purpose of this study is to compare visual improvement and total number of intraocular injections in eyes with macular edema following central retinal vein occlusion (CRVO)after initial treatment with Ozurdex (dexamethasone implant) or Avastin (bevacizumab).

ELIGIBILITY:
Inclusion Criteria:

* Presence of central retinal vein occlusion (CRVO)
* Age 18 years or older
* ETDRS (Early Treatment Diabetic Retinopathy Study) Visual acuity between 3 and 72 letters and approximate Snellen equivalent of 20/40 to 20/800
* OCT Central foveal thickness >250 microns
* Negative pregnancy test for women of childbearing potential
* Ability to provide written informed consent
* Capable of complying with study protocol

Exclusion Criteria:

* History of glaucoma in the study eye with intraocular pressure >21mmHg on more than one topical medication. Combination drugs are considered more than one medication
* History of steroid-related glaucoma (steroid response)
* Previous intraocular injection of steroid medication within 90 days
* Avastin (bevacizumab) or Lucentis (ranibizumab) within 60 days
* Evidence of significant retinal ischemia on fluorescein angiography in the opinion of the treating physician
* Previous intraocular surgery (e.g. Cataract Surgery) with in 60 days
* Concurrent ocular disease that would limit visual acuity in the opinion of the treating physician
* Dense cataract that precludes clinical examination and retinal imaging of the retina
* History of allergy to dexamethasone, bevacizumab, betadine
* Ocular or systemic conditions that may pose a threat to the health of the subject in the opinion of the treating physician
* Unwilling or unable to follow or comply with all study related procedures
* Current participation in another clinical medical investigation or trial or has received any investigational drug within 12 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent A Deramo, M.D, Principal Investigator — Long Island Vitreoretinal Consultants
Locations (4):
- United States (4):
  - Retina Vitreous Center, Toms River, New Jersey
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Long Island Vitreoretinal Consultants, Hauppauge, New York
  - Long Island Vitreoretinal Consultants, Riverhead, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozurdex & Avastin: Subjects randomized to this arm will receive one initial treatment with Ozurdex then treated with Avastin if needed.
  Ozurdex: Ozurdex, 0.7mg dexamethasone
  Avastin: Formulated as a 1.25mg/0.05ml sterile solution given by intravitreal injection monthly as needed.
- Avastin Only: Subjects randomized to this arm will receive one initial treatment with Avastin then treated with Avastin if needed.
  Avastin: Formulated as a 1.25mg/0.05ml sterile solution given by intravitreal injection monthly as needed.
Period: Overall Study
Arm/Group | Ozurdex & Avastin | Avastin Only
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 9 | 10 | 19
Age, Continuous [Mean (Full Range); unit: years] | 68.8 [43 to 92] | 74.3 [62 to 86] | 71.3 [43 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Change in Visual Acuity (Number of ETDRS Early Treatment Diabetic Retinopathy Study Letters), at Month 6 as Compared With Baseline in Each Treatment Arm
Description: The change in visual acuity (number of ETDRS - Early Treatment Diabetic Retinopathy Study letters), at Month 6 as compared with baseline in each treatment arm
Time Frame: Baseline - Month 6
Measure: Mean (Full Range); unit: Letters Gain/Loss
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 13
Letters Gain/Loss | 11.1 [-7 to 38] | 16.1 [-2 to 39]

2. Primary Outcome: The Total Number of Additional Avastin Injections Following Initial Treatment in Each Treatment Arm
Description: Total Number of addiitonal Avastin injections during study- From baseline to Month 6
Time Frame: Baseline - Month 6
Measure: Mean (Full Range); unit: Injections
Arm/Group | Ozurdex & Avastin | Avastin Only
Number analyzed (Participants) | 14 | 13
Injections | 2.5 [1 to 6] | 5.1 [3 to 6]

3. Secondary Outcome: Change in Central Mean Thickness Based on OCT
Description: Change in Central Mean Thickness based on OCT from baseline to Month 6t
Time Frame: Baseline to 6 Months
Measure: Mean (Full Range); unit: Microns on OCT
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 13
Microns on OCT
  Initial OCT Measure at Basline | 703 [344 to 1255] | 790 [496 to 1183]
  Final OCT measure at Month 6 | 353 [189 to 605] | 408 [149 to 710]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the study period of 6 months.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes